CLINICAL TRIAL: NCT04144127
Title: A Soccer-based Lifestyle Intervention vs mHealth-based Physical Activity Intervention to Improve Bone Health and Metabolic Health in Prostate Cancer Survivors
Brief Title: Soccer Intervention in Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberto Felipe Lobelo, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00110890; P30CA138292 (NIH)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soccer Group (Experimental): Participants in the soccer group will participate in soccer drills and other fitness routines (two 1-hour sessions per week). They will meet with the soccer coach after the soccer sessions to discuss the lifestyle education topics (Life's Simple 7 education topics). During the soccer sessions participants will be fitted with a wearable soccer-specific device to measure how much they move and their heart rate. All participants will receive a Garmin Vivofit wearable device to help monitor their PA goals and achievements.
  Interventions: Behavioral: Soccer

INTERVENTIONS:
Behavioral: Soccer — * Soccer drills and other fitness routines (two 1-hour sessions per week)
  * In person education in Life's Simple 7 to help improve life through Lifestyle changes: smoking status, physical activity, weight, diet, blood glucose, cholesterol, and blood pressure.
  Other Names: Recreational Soccer (RS)

SUMMARY:
This study seeks to directly test the implementation feasibility of a soccer-based and lifestyle education intervention to determine the effects on bone health, body composition, mental health, functional and cardiometabolic status among prostate cancer survivors.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common cancer in men in the U.S. and in other industrialized countries. The lifetime probability of PCa in males is one in nine, and it has a high economic burden, with costs expected to rise. Modern tailored treatment approaches, including androgen deprivation therapy (ADT), have resulted in longer life expectancy, but also longer treatment periods, which lead to significant adverse side effects. These often include decreased bone mineral density (BMD), increased risk of fractures, low functional capacity, loss of lean body mass (LBM), increased fat mass, insulin resistance, psychological distress and pain. Of particular concern is a sharp decline in bone health, with systemic bone loss caused by PCa-produced osteoclastogenic cytokines and drug interventions. Independent of disease stage, fractures in PCa patients are predictors of survival. In addition, concomitant physical inactivity and stress during and after treatment predispose PCa patients to elevated risk of deconditioning, BMD loss, cardiovascular and metabolic disease morbidity and mortality.

Exercise-based lifestyle interventions aimed at counteracting treatment-induced adverse effects have been shown to be safe and effective in improving bone, functional and cardiometabolic health for patients with PCa. However, men, in general, are harder to engage in physical activity (PA) and lifestyle interventions. As an alternative to traditional exercise programs, recreational team sports provide a unique environment that may lead to increased physical activity participation and motivation to engage in other lifestyle changes. More than any other sport, recreational soccer (RS) has been shown to be a successful health intervention in patients with, or at risk of chronic diseases, including PCa.

Leveraging the growing enthusiasm around soccer in Atlanta and the U.S. may lead to increased interest, participation, retention and engagement in lifestyle change programming among PCa survivors. Therefore, this study seeks to directly test the implementation feasibility of a soccer-based lifestyle change intervention to determine the effect on bone health, body composition, mental health, functional and cardiometabolic status among PCa survivors.

Participants will be offered an intensive intervention including RS programming and lifestyle education. The group will receive RS, consisting of conditioning drills and games, adapted to the population during 60-minute sessions twice per week. The researchers will evaluate health outcomes at baseline and after 3 months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. men aged 18-79 years
2. PCa survivors that had at least 6 months of hormone therapy (i.e. ADT with testosterone lowering agents) within the past 10 years
3. not engaged in soccer practice or other exercise or lifestyle intervention program for the past 12 months
4. availability of smartphone to receive text messages
5. treating Oncologist clearance
6. ability to read in English or Spanish and provide informed consent

Exclusion Criteria:

1. BMI > 40 kg/m^2
2. resting BP ≥170/100 at screening or uncontrolled hypertension
3. any mobility issues or exercise program contraindications
4. a recent (i.e., within 12 months) myocardial infarction, diagnosis of congestive heart disease, other active cancer
5. bone or organ metastases
6. chemotherapy within past 6 months
7. therapies and diseases of bone unrelated to PCa e.g. systemic glucocorticoids, bisphosphonates, teriparatide, denosumab, osteomalacia; osteosarcoma; Paget's disease; systemic lupus erythematosus; inflammatory bowel diseases, rheumatoid arthritis; thyroid/parathyroid disorder or mental illness
8. not coronavirus disease 2019 (COVID-19) vaccinated

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Felipe Lobelo, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Soccer Group: Participants in the soccer group will participate in soccer drills and other fitness routines (two 1-hour sessions per week). They will meet with the soccer coach after the soccer sessions to discuss the lifestyle education topics (Life's Simple 7 education topics). During the soccer sessions participants will be fitted with a wearable soccer-specific device to measure how much they move and their heart rate. All participants will receive a Garmin Vivofit wearable device to help monitor their PA goals and achievements.
  Soccer: - Soccer drills and other fitness routines (two 1-hour sessions per week)
  - In person education in Life's Simple 7 to help improve life through Lifestyle changes: smoking status, physical activity, weight, diet, blood glucose, cholesterol, and blood pressure.
Period: Overall Study
Arm/Group | Soccer Group
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density (BMD)
Description: Bone mineral density will be measured by dual x-ray absorptiometry (DXA) scan at the lumbar spine (L2-L4). Decreased BMD a is associated with an increased risk of fractures.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
mg/cm^3
  Baseline | 1.2 (0.3)
  3 months post-intervention | 1.2 (0.3)

2. Secondary Outcome: Total Hip BMD
Description: Bone mineral density will be measured by dual x-ray absorptiometry (DXA) scan at the hip. Decreased BMD a is associated with an increased risk of fractures.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
mg/cm^3
  Baseline | 1.2 (0.1)
  3 months post-intervention | 1.2 (0.1)

3. Secondary Outcome: Osteocalcin Level
Description: Osteocalcin is marker of bone formation. The normal range for osteocalcin varies by lab and elevated levels are seen in patients with bone diseases characterized by increased bone turnover.
Time Frame: Baseline, 3 months post-intervention
Population: Unable to collect sample for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

4. Secondary Outcome: C-terminal Telopeptide of Collagen (CTx)
Description: C-terminal telopeptide of collagen (CTx) is a bone resorption marker. Increased levels indicate increased bone resorption with conditions such as osteoporosis and osteopenia.
Time Frame: Baseline, 3 months post-intervention
Population: Unable to collect information for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Weight
Description: Weight is measured in kilograms (kg).
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
Kg
  Baseline | 111.6 (10.4)
  3 months post-intervention | 106.6 (11.1)

6. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI) is weight in kilograms divided by the square of height in meters.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
kg/m^2
  Baseline | 34.1 (1.7)
  3 months post-intervention | 32.7 (2.0)

7. Secondary Outcome: Percentage of Body Fat
Description: Body fat is measured by dual x-ray absorptiometry (DXA) scan.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: % of body fat
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
% of body fat
  Baseline | 42.1 (3.3)
  3 months post-intervention | 40.9 (2.9)

8. Secondary Outcome: Waist Circumference
Description: Waist circumference is measured in centimeters (cm).
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: cms
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
cms
  Baseline | 120.6 (0.5)
  3 months post-intervention | 117.3 (0.5)

9. Secondary Outcome: Lean Body Mass
Description: Lean body mass is body weight minus weight from body fat.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
lbs
  Baseline | 138.9 (16.9)
  3 months post-intervention | 135.7 (17.9)

10. Secondary Outcome: Resting Heart Rate
Description: The normal resting heart rate in adults is between 60 and 100 beats per minute (bpm). A lower resting heart rate indicates that the person has better fitness as the heart is working more efficiently.
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

11. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (BP) will be measured while sitting using a calibrated electronic blood pressure sphygmomanometer at Baseline and at 3 months post-intervention. A normal systolic blood pressure reading is lower than 120 mmHg. BP values higher than 120 mmHg correlate with worse outcome.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
mmHg
  Baseline | 140.3 (15.9)
  3 months post-intervention | 126.3 (22.3)

12. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure (BP) will be measured while sitting using a calibrated electronic blood pressure sphygmomanometer prior to any activity (Baseline) and at 3 months post-intervention. A normal diastolic blood pressure reading is lower than 80 mmHg. BP values higher than 80 mmHg correlate with worse outcome.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
mmHg
  Baseline | 79 (12.5)
  3 months post-intervention | 68.3 (11.9)

13. Secondary Outcome: Aerobic Capacity
Description: Aerobic capacity is measured by 6 minute walk test distance (meters).
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
meters
  Baseline | 536.7 (80.8)
  3 months post-intervention | 497.7 (54.1)

14. Secondary Outcome: Muscle Strength
Description: Muscle strength is measured as hand grip strength (kg). Hand grip was measured using a study approved dynamometer to test the maximum isometric strength of the hand and forearm muscles of the dominant hand. An increase in values means that grip strength is improving.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
Kg
  Baseline | 36.1 (4.3)
  3 months post-intervention | 37.7 (4.4)

15. Secondary Outcome: Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) Score
Description: Physical activity self-efficacy is assessed with the BREQ-2 instrument. The BREQ-2 has 19 items measuring motivation to exercise, with 5 motivational styles examined: intrinsic regulation (the respondent finds physical activity enjoyable), identified regulation (the respondent sees benefits of physical activity), introjected regulation (physical activity is done to increase self-esteem or avoid negative feelings with not performing exercise), external regulation (physical activity is done based on rewards or punishments from someone else), and amotivation (the respondent has no motivation to engage in physical activity). Responses are given on a 5 point Likert scale where 0=not true for me, and 4=very true for me. A relative autonomy index (RAI) can be calculated by weighting the scores for each motivational style factor. The weights range from 3 to -3 and total RAI scores range from -24 to 20. Higher scores indicate greater self-determined motivation to engage in physical activity.
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

16. Secondary Outcome: Dietary Intake
Description: The dietary intake is measured using the Nutrition Database System for Research (NDSR) 24-hour dietary recall. The NDSR is a dietary analysis software application used to collect and calculate nutritional intake.
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants Smoking Cigarettes
Description: Smoking habits are assessed with the National Health and Nutrition Examination Survey (NHANES) 2019-2020 for smoking and tobacco use. This instrument includes 24 items and the number of questions that a respondent answers depends on their past and current smoking behaviors. Participants are asked if they currently smoke cigarettes and possible responses are: "every day", "some days", and "not at all".
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

18. Secondary Outcome: Alcohol Habits
Description: Number of alcohol beverages per week will be recorded.
Time Frame: Baseline, 3 months post-intervention
Population: Information for this outcome was not collected.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

19. Secondary Outcome: Sleep Time
Description: Average sleep time will be collected in minutes per day.
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

20. Secondary Outcome: Weekly Steps
Description: Participants will be asked to wear a Garmin fitness tracker throughout the study and physical activity will be measured as steps taken per week.
Time Frame: Baseline, 3 months post-intervention
Population: Information was not collected for this study outcome.
Arm/Group | Soccer Group
Number analyzed (Participants) | 0

21. Secondary Outcome: SF-12 Health Survey Score
Description: Quality of life is assessed with the SF-12 Health Survey. The SF-12 is a multipurpose, standardized self-report short form survey with 12 questions assessing mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for each component ranging from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
score on a scale
  Baseline PCS | 44.2 (17.4)
  3 months post-intervention PCS | 47.2 (9.5)
  Baseline MCS | 53.2 (8.7)
  3 months post-intervention MCS | 53.6 (4.9)

22. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CESD) Score
Description: Symptoms of depression are assessed with the CESD. The CESD is a 20-item questionnaire asking about feelings and behaviors during the past week. Responses are given on a 4-point scale where 0 = rarely or none of the time (less than 1 day), 1 = some or a little of the time (1-2 days), 2 = occasionally or a moderate amount of time (3-4 days), and 3 = most or all of the time (5-7 days). Scores range from 0 to 60 with high scores indicating greater depressive symptoms.
Time Frame: Baseline, 3 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soccer Group
Number analyzed (Participants) | 3
score on a scale
  Baseline | 4.3 (5.9)
  3 months post-intervention | 5.3 (5.9)

ADVERSE EVENTS:
Time Frame: Up to 3 months post-intervention.
Arm/Group | Soccer Group
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04144127/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04144127/ICF_000.pdf